CLINICAL TRIAL: NCT06762288
Title: Analgesic Effectiveness Of Ultrasound-Guided Transversus Abdominis Plan (TAP) Block In Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Transversus Abdominis Plan (TAP) Block In Transcatheter Aortic Valve Implantation (TAVI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kerem Erkalp, MD, Prof, professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia; Analgesia; Block; Aortic Valve Stenosis
Keywords: transversus abdominis plan block; tavi; transcatheter aortic valve implantation; nerve block; aortic stenosis; interventional cardiology; anesthesia; ultrasound
MeSH Terms: conditions — Agnosia; Bites and Stings; Aortic Valve Stenosis | interventions — Ultrasonography; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Local anesthesia and sedation will be applied as standard procedure and unilateral USG-guided TAP block will be performed. In both groups, an additional dose of anesthetic drugs (midazolam 0.05mg/kg and fentanyl 1mcg/kg or propofol 0.5-1mg/kg) will be administered slowly IV when the patient feels pain, wakes up (BIS>80) or moves.
  Interventions: Device: Ultrasound; Procedure: Local anesthesia and sedation
- Control group (Sham Comparator): Local anesthesia and sedation will be applied as standard procedure in the control group (C) (n: 25). In both groups, an additional dose of anesthetic drugs (midazolam 0.05mg/kg and fentanyl 1mcg/kg or propofol 0.5-1mg/kg or ) will be administered slowly IV when the patient feels pain, wakes up (BIS>80) or moves
  Interventions: Procedure: Local anesthesia and sedation

INTERVENTIONS:
Device: Ultrasound — Sedation and local anesthesia to the surgical field will be applied as standard procedure and unilateral USG-guided TAP block will be performed to the patients who will undergo TAVİ.
  Arms: Block group
Procedure: Local anesthesia and sedation — Sedation and local anesthesia to the surgical field will be applied to the patients who will undergo TAVİ.

SUMMARY:
Hemodynamic stability is the main goal of the anesthetic method during TAVI. Pain during the procedure may cause patients to move therefore hemodynamic instability. This may lead to undesirable complications for the patient and the physician. At the same time, it may affect the process quality and cause the processing time to be extended. In this prospective-randomised study, ultrasound-guided transversus abdominis plan block will be performed to reduce pain. We aimed to contribute to the reduction of undesirable outcomes for the patient and physician by providing adequate anesthesia with TAP block accompanied by sedation, and to present its impact on the quality of the healthcare service provided by evaluating patient and physician satisfaction.

DETAILED DESCRIPTION:
While common aortic valve stenosis was previously treated with surgical aortic valve replacement, with the developments in the field of interventional cardiology, TAVI has emerged as an alternative to surgery in recent years and has become the first choice in the treatment of inoperable patients with severe aortic stenosis. Especially patients who are elderly, have chronic illnesses, have a high surgical risk, and whose general health condition is not suitable for surgery can be treated with this method.

Mostly the femoral artery is preferred for TAVİ access because it has a large lumen (8-9 mm) and has less anatomical variation. After the inguinal ligament, the iliac artery, originating from the abdominal aorta, is called the femoral artery. Since this region is safe, it is preferred in cardiac interventions.

Transversus abdominis plane (TAP) block aims to block the ilioinguinal and iliohypogastric nerves which contribute to the sensory innervation of the femoral region used for endovascular cardiac interventions. No studies have been found on the analgesic efficacy of TAP block in TAVİ procedures.

Local anesthesia and sedation as standard procedure will be applied to the control group (C) (n: 25). In TAP block group (TAP) (n:25) standard procedure and unilateral USG-guided TAP block will be performed. In both groups, an additional dose of anesthetic drugs (midazolam 0.05mg/kg and fentanyl 1mcg/kg or propofol 0.5-1mg/kg) will be administered slowly IV when the patient feels pain, wakes up (BIS>80) or moves.

Patients' demographic data, hemodynamic parameters, total anesthetic drug consumption, procedure duration, complications seen during the procedure will be recorded. The highest pain level felt during procedure, when placing and withdrawing sheath and 4 hours after removal will be recorded according to the Numeric rating scale-11 (NRS-11) scoring system. 5-point Likert scale will be used for patient and physician satisfaction.

Cardiac endovascular catheterization procedures such as TAVI are often anxiety-provoking and uncomfortable for patients. The anesthesia method may vary depending on the experience of the cardiology team, the characteristics of the patients and the procedure to be performed. In TAVI procedures, which were initially performed under general anesthesia, a combination of local anesthesia and sedation was preferred as the team's experience developed. Hemodynamic stability and patient immobilization are the main goals of the anesthetic method during TAVI. Due to pain, patients may develop hemodynamic instability and may move. This is an undesirable situation for cardiac patients. It may affect the quality of the procedure for the cardiologist and may cause complications and longer procedure times. Examining the effectiveness of anesthesia by applying TAP block accompanied by sedation and physician and patient satisfaction during and after the procedure forms the basis of the research. First aim of the study is to demonstrate the analgesic effectiveness of ultrasound-guided TAP block application in the femoral region before the procedure in 50 patients who underwent TAVI. Secondary aims are to reduce the need for anesthetic drugs and to investigate patient and physician satisfaction during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* TAVI procedures
* over 18 years of age
* INR < 1,5
* elective procedures
* Signing the volunteer consent form
* Providing optimal images in ultrasound imaging

Exclusion Criteria:

* < 18 yers of age
* emergency procedures
* morbidly obese patients (BMI>35kg/m2)
* Advanced decompensated heart failure with New york Heart Association (NYHA) stage 4
* Those who have skin infection, lesion, hematoma in the area to be blocked
* Cannot be communicated and cannot be given a position
* Allergic to the prescribed medications
* Pregnants
* Those who refused to sign volunteer consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The pain assessed by the Numeric Rating Scale-11 (NRS-11) to measure the analgesic efficacy of TAP | 6 months
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable

SECONDARY OUTCOMES:
Investigation patient and physician satisfaction assessed by 5-point Likert scale | 6 months
  A 5-point Likert scale is a psychometric response method where respondents can easily answer questions and state their level of agreement in five points. The 5-point Likert scale consists of the below points - (1) Strongly Disagree; (2) Disagree; (3) Neither Agree nor Disagree; (4) Agree; (5) Strongly Agree.For both patients and physicians satisfaction 5-point Likert scale will be used.
Evaluate the need for anesthetic drugs | 6 months
  reduction of the need for anesthetic drugs with tap block

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, professor, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No